CLINICAL TRIAL: NCT02536833
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, and Efficacy of SM04690 Injected in the Target Knee Joint of Moderately to Severely Symptomatic Osteoarthritis Subjects
Brief Title: A Study Evaluating the Safety, Tolerability, and Efficacy of SM04690 Injected in the Target Knee Joint of Moderately to Severely Symptomatic Osteoarthritis Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SM04690-OA-02
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Samumed; SM04690
MeSH Terms: conditions — Osteoarthritis | interventions — lorecivivint

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 0.03 mg SM04690 (Experimental): Single intra-articular injection of SM04690 0.03 mg in 2 mL injectable suspension
  Interventions: Drug: SM04690
- 0.07 mg SM04690 (Experimental): Single intra-articular injection of SM04690 0.07 mg in 2 mL injectable suspension
  Interventions: Drug: SM04690
- 0.23 mg SM04690 (Experimental): Single intra-articular injection of SM04690 0.23 mg in 2 mL injectable suspension
  Interventions: Drug: SM04690
- Placebo (Placebo Comparator): Single intra-articular injection of SM04690 0 mg in 2 mL phosphate buffered saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SM04690
  Arms: 0.03 mg SM04690; 0.07 mg SM04690; 0.23 mg SM04690
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy, safety, and tolerability of three different strengths of SM04690 injected in the target knee joint of moderately to severely symptomatic osteoarthritis (OA) subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 40 and 80 years of age, inclusive, in general good health
2. Ambulatory (single assistive devices such as canes allowed if needed less than 50% of the time, subjects requiring a walker are excluded)
3. Established diagnosis of primary femorotibial OA in the target knee by standard American College of Rheumatology (ACR) criteria for at least 6 months (clinical AND radiographic criteria); if bilateral knee OA is present, the target knee is defined as the knee with greater pain at screening based on the subject's evaluation and the Investigator's clinical judgment
4. Radiographic disease Stage 2 or 3 in the target knee according to the Kellgren-Lawrence grading of knee OA as assessed by independent central readers
5. Screening pain visual analog scale (VAS) score of 30-80 mm (on a scale of 0-100 mm) for the target knee while on symptomatic oral treatment at screening (if the subject requires oral treatment)
6. Total WOMAC score of 72-192 (out of 240) for the target knee while on symptomatic oral treatment at screening (if the subject requires oral treatment)
7. Willingness to omit the following for 24 hours prior to all Study Visits, excluding the Screening Visit:

   1. Pain medications
   2. Medications or supplements for the treatment of OA
   3. Participation in a formalized in-office and/or supervised OA disease program (e.g., a prescribed patient education program, physiotherapy, etc.)
8. Full understanding of the requirements of the study and willingness to comply with all study visits and assessments
9. Subjects must have read and understood the informed consent form, and must have signed it prior to any study-related procedure being performed
10. Subject's Day 1 visit must occur while enrollment into the study is open

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Women of childbearing potential (i.e., who are not surgically sterile or postmenopausal as defined by no menstrual periods for 12 consecutive months and no other biological or physiological cause for amenorrhea can be identified); males who are sexually active and have a partner who is capable of becoming pregnant, neither of which have had surgery to become sterilized, who are not using an effective method of birth control (e.g., surgically-implanted hormonal therapy, intrauterine devices or oral birth control with barrier method)
3. Body mass index (BMI) >40
4. Partial or complete joint replacement in the target knee
5. Previous exposure to SM04690
6. Major surgery (e.g., interventional arthroscopy) in the target knee within 52 weeks prior to any study injection
7. Any planned or elective surgery during the study period
8. Significant and clinically evident misalignment of the target knee that would impact subject function, as determined by the Investigator
9. History of malignancy within the last 5 years; however, subjects with prior history of in situ cancer or basal or squamous cell skin cancer are eligible. Subjects with other malignancies are eligible if they have been continuously disease free for at least 5 years prior to any study injection
10. Clinically significant abnormal Screening Visit hematology values, blood chemistry values, HbA1c, or urinalysis values as determined by the investigator
11. Any condition, including laboratory findings (not included in the Screening Visit laboratory tests) and findings in the medical history or in the pre-study assessments, that, in the opinion of the Investigator, constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
12. Comorbid conditions that could affect pain assessment of the target knee, including, but not limited to, inflammatory rheumatic conditions such as rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, diabetic neuropathy, pseudogout, gout, and fibromyalgia
13. Other conditions that, in the opinion of the Investigator, could affect pain assessment of the target knee, including, but not limited to, symptomatic hip osteoarthritis and symptomatic degenerative disc disease
14. Any diagnosed psychiatric condition that includes, but is not limited to, a history of mania, bipolar disorder, psychotic disorder, schizophrenia, major depressive disorder, or generalized anxiety disorder
15. Participation in a clinical research trial that included the receipt of an investigational product or any experimental therapeutic procedure within 12 weeks prior to any study injection; the last date of participation in the trial, not the last date of receipt of investigational product, must be at least 12 weeks prior to Study Visit Day 1
16. Treatment of the target knee with systemic or intra-articular corticosteroids (e.g., methylprednisolone) within 8 weeks prior to Study Visit Day 1
17. Viscosupplementation (e.g., hyaluronic acid) in the target knee within 24 weeks prior to Study Visit Day 1
18. Effusion of the target knee clinically requiring aspiration within 12 weeks prior to Study Visit Day 1
19. Use of electrotherapy, acupuncture, and/or chiropractic treatments for knee OA within 4 weeks prior to Study Visit Day 1
20. Any known active infections, including suspicion of intra-articular infection, hepatitis B or hepatitis C infection, and/or infections that may compromise the immune system such as human immunodeficiency virus (HIV)
21. Subjects taking prescription medications for OA who have not maintained a stable therapeutic regimen for a minimum of 12 weeks prior to Study Visit Day 1
22. Subjects requiring the chronic use (i.e., regular and consistent use for ≥ 12 weeks) of the medications listed below within 12 weeks prior to Study Visit Day 1:

    1. Opioids, both oral (e.g., tramadol) or transdermal (e.g., fentanyl patches) formulations
    2. Centrally acting analgesics (e.g., duloxetine)
    3. Glucocorticoids (e.g., methylprednisolone) administered by any route, with exception of inhaled, intranasal, and ophthalmic solutions
23. Any chronic condition that has not been well controlled or subjects with a chronic condition who have not maintained a stable therapeutic regimen of a prescription therapy for a minimum of 12 weeks prior to Study Visit Day 1. In addition, the following subjects will be excluded:

    1. Subjects with a baseline HbA1c >9
    2. Subjects with uncontrolled hypertension in the opinion of the investigator
    3. Subjects with symptomatic coronary artery disease in the opinion of the investigator
24. Subjects who have a current or pending disability claim, workers' compensation, or litigation(s) that may compromise response to treatment
25. Subjects who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at the investigative site, or are directly affiliated with the study at the investigative site
26. Subjects employed by Samumed, LLC, or any of its affiliates or development partners (that is, an employee, temporary contract worker, or designee) responsible for the conduct of the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (36):
- United States (36):
  - Research Site, Mobile, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, El Cajon, California
  - Research Site, Rancho Mirage, California
  - Research Site, Spring Valley, California
  - Research Site, Denver, Colorado
  - Research Site, Clearwater, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Woodstock, Georgia
  - Research Site, Newton, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Frederick, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site 1, St Louis, Missouri
  - Research Site 2, St Louis, Missouri
  - Research Site, Orchard Park, New York
  - Research Site, Rochester, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Knoxville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, West Layton, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Franklin, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yazici Y, McAlindon TE, Gibofsky A, Lane NE, Clauw D, Jones M, Bergfeld J, Swearingen CJ, DiFrancesco A, Simsek I, Tambiah J, Hochberg MC. Lorecivivint, a Novel Intraarticular CDC-like Kinase 2 and Dual-Specificity Tyrosine Phosphorylation-Regulated Kinase 1A Inhibitor and Wnt Pathway Modulator for the Treatment of Knee Osteoarthritis: A Phase II Randomized Trial. Arthritis Rheumatol. 2020 Oct;72(10):1694-1706. doi: 10.1002/art.41315. Epub 2020 Sep 6. PMID 32432388
- [Derived] Tambiah J, Kennedy S, Swearingen C, McAlindon T, Yazici Y. Impact of structural severity on outcomes in knee osteoarthritis: an analysis of data from phase 2 and phase 3 lorecivivint clinical trials. Rheumatology (Oxford). 2025 May 1;64(5):2583-2590. doi: 10.1093/rheumatology/keae610. PMID 39495154

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo
Started | 112 | 117 | 110 | 116
Completed | 103 | 107 | 95 | 97
Not Completed | 9 | 10 | 15 | 19
Not completed — Discontinued Before Treatment | 0 | 0 | 1 | 2
Not completed — Adverse Event | 1 | 3 | 4 | 1
Not completed — Lost to Follow-up | 2 | 1 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Site Terminated by Sponsor | 2 | 2 | 2 | 2
Not completed — Subject Non-Compliance | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3 | 5 | 11

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population is the Intent-to-Treat (ITT) Analysis Set (i.e. all participants who were randomized).
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo | Total
Number analyzed (Participants) | 112 | 117 | 110 | 116 | 455
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (9) | 60 (8.2) | 61.3 (8.7) | 60.7 (8.9) | 60.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 60 | 68 | 72 | 268
  Male | 44 | 57 | 42 | 44 | 187
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 23 | 17 | 21 | 81
  Not Hispanic or Latino | 92 | 94 | 93 | 95 | 374
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 2 | 3
  Asian | 1 | 0 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 18 | 14 | 12 | 10 | 54
  White | 92 | 102 | 96 | 102 | 392
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Kellgren-Lawrence Grade [Count of Participants; unit: Participants] — Participants' knee osteoarthritis was graded in accordance with the following definitions of Kellgren-Lawrence Grade: None (Grade 0) - Normal appearance of the knee; Doubtful (Grade 1): Doubtful narrowing of joint space and possible osteophytic lipping; Minimal (Grade 2): Definite osteophytes and possible narrowing of joint space; Moderate (Grade 3): Moderate multiple osteophytes, definite narrowing of the joint space, some sclerosis and possible deformity of bone ends; Severe (Grade 4): Large osteophytes, marked narrowing of joint space, severe sclerosis and definite deformity of bone ends.
  Participants
    Grade 2 | 38 | 43 | 39 | 41 | 161
    Grade 3 | 74 | 74 | 70 | 74 | 292
    Grade 4 | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Osteoarthritis (OA) Pain in the Target Knee
Description: Change from baseline OA pain in the target knee as assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Numeric Rating Scale (NRS 3.1) pain subscore (WOMAC Pain) at Week 13. The WOMAC is a widely-used, proprietary outcome measurement tool used by health professionals to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Pain subscore is reported ranging from 0 to 100.
Time Frame: Baseline and Week 13
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo
Number analyzed (Participants) | 112 | 117 | 110 | 116
score on a scale | -23.3 (2.2) | -23.5 (2.1) | -21.3 (2.2) | -22.1 (2.1)
Statistical Analysis 1: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.575, ANCOVA; Mean Difference (Final Values) = -1.46, 95% CI 2-sided [-6.57 to 3.65]
Statistical Analysis 2: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.643, ANCOVA; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-6.63 to 4.09]
Statistical Analysis 3: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.901, ANCOVA; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-5.07 to 5.75]

2. Secondary Outcome: Change From Baseline OA Pain in the Target Knee
Description: Change from baseline OA pain in the target knee as assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Numeric Rating Scale (NRS 3.1) pain subscore (WOMAC Pain) at Week 26. The WOMAC is a widely-used, proprietary outcome measurement tool used by health professionals to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Pain subscore is reported ranging from 0 to 100.
Time Frame: Baseline and Week 26
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo
Number analyzed (Participants) | 112 | 117 | 110 | 116
score on a scale | -24.7 (2.3) | -27.3 (2.0) | -23.3 (2.1) | -24.4 (2.1)
Statistical Analysis 1: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.271, ANCOVA; Mean Difference (Final Values) = -2.99, 95% CI 2-sided [-8.31 to 2.33]
Statistical Analysis 2: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.898, ANCOVA; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-6.06 to 5.32]
Statistical Analysis 3: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.795, ANCOVA; Mean Difference (Final Values) = 0.72, 95% CI 2-sided [-4.74 to 6.18]

3. Secondary Outcome: Change From Baseline OA Function in the Target Knee
Description: Change from baseline OA function in the target knee as assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Numeric Rating Scale (NRS 3.1) physical functioning subscore (WOMAC Function) at Week 13. The WOMAC is a widely-used, proprietary outcome measurement tool used by health professionals to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Function subscore is reported ranging from 0 to 100.
Time Frame: Baseline and Week 13
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo
Number analyzed (Participants) | 112 | 117 | 110 | 116
score on a scale | -24.5 (2.1) | -26.3 (2.0) | -22.6 (2.1) | -22.8 (2.1)
Statistical Analysis 1: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.283, ANCOVA; Mean Difference (Final Values) = -2.74, 95% CI 2-sided [-7.74 to 2.26]
Statistical Analysis 2: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.588, ANCOVA; Mean Difference (Final Values) = -1.48, 95% CI 2-sided [-6.82 to 3.86]
Statistical Analysis 3: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.853, ANCOVA; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-5.76 to 4.76]

4. Secondary Outcome: Change From Baseline OA Function in the Target Knee
Description: Change from baseline OA function in the target knee as assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Numeric Rating Scale (NRS 3.1) physical functioning subscore (WOMAC Function) at Week 26. The WOMAC is a widely-used, proprietary outcome measurement tool used by health professionals to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Function subscore is reported ranging from 0 to 100.
Time Frame: Baseline and Week 26
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo
Number analyzed (Participants) | 112 | 117 | 110 | 116
score on a scale | -25.1 (2.2) | -28.6 (2.0) | -24.1 (2.0) | -25.1 (2.1)
Statistical Analysis 1: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.292, ANCOVA; Mean Difference (Final Values) = -2.89, 95% CI 2-sided [-8.26 to 2.49]
Statistical Analysis 2: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.931, ANCOVA; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-5.34 to 5.83]
Statistical Analysis 3: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.878, ANCOVA; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-4.92 to 5.76]

5. Secondary Outcome: Change From Baseline OA Disease Activity as Assessed by the Patient
Description: Change from baseline OA disease activity as assessed by the Patient Global Assessment at Week 13. The Patient Global Assessment was completed using a 100 mm visual analog scale (VAS) adapted from the Patient Assessment Form © 1999, American College of Rheumatology. The subject rated how well he/she was doing, considering all the ways in which illness and health conditions may affected him/her. The VAS scale was anchored by "Very Well" on the left (scored as 0) and "Very Poorly" on the right (scored as 100). Higher scores indicated poorer disease assessment by the subject.
Time Frame: Baseline and Week 13
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo
Number analyzed (Participants) | 112 | 117 | 110 | 116
mm | -18.1 (2.3) | -13.7 (2.3) | -14.6 (2.6) | -14.0 (2.3)
Statistical Analysis 1: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.648, ANCOVA; Mean Difference (Final Values) = 1.16, 95% CI 2-sided [-3.83 to 6.16]
Statistical Analysis 2: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.209, ANCOVA; Mean Difference (Final Values) = -3.14, 95% CI 2-sided [-8.02 to 1.75]
Statistical Analysis 3: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.915, ANCOVA; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-4.78 to 5.33]

6. Secondary Outcome: Change From Baseline OA Disease Activity as Assessed by the Patient
Description: Change from baseline OA disease activity as assessed by the Patient Global Assessment at Week 26. The Patient Global Assessment was completed using a 100 mm visual analog scale (VAS) adapted from the Patient Assessment Form © 1999, American College of Rheumatology. The subject rated how well he/she was doing, considering all the ways in which illness and health conditions may affected him/her. The VAS scale was anchored by "Very Well" on the left (scored as 0) and "Very Poorly" on the right (scored as 100). Higher scores indicated poorer disease assessment by the subject.
Time Frame: Baseline and Week 26
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo
Number analyzed (Participants) | 112 | 117 | 110 | 116
score on a scale | -21.3 (2.4) | -17.5 (2.3) | -17.2 (2.6) | -16.6 (2.6)
Statistical Analysis 1: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.969, ANCOVA; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-5.16 to 5.36]
Statistical Analysis 2: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.174, ANCOVA; Mean Difference (Final Values) = -3.64, 95% CI 2-sided [-8.89 to 1.61]
Statistical Analysis 3: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.908, ANCOVA; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-4.97 to 5.59]

7. Secondary Outcome: Change From Baseline in Medial Joint Space Width of Target Knee
Description: Change from baseline in medial joint space width as documented by X-ray of the target knee at Week 26.
Time Frame: Baseline and Week 26
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo
Number analyzed (Participants) | 112 | 117 | 110 | 116
mm | -0.07 (0.06) | -0.11 (0.08) | -0.02 (0.06) | -0.20 (0.06)
Statistical Analysis 1: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.334, ANCOVA; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.10 to 0.29]
Statistical Analysis 2: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.124, ANCOVA; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.04 to 0.30]
Statistical Analysis 3: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.032, ANCOVA; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [0.02 to 0.36]

8. Other Pre Specified Outcome: Change From Baseline OA Pain in the Target Knee
Description: Change from baseline OA pain in the target knee as assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Numeric Rating Scale (NRS 3.1) pain subscore (WOMAC Pain) at Week 52. The WOMAC is a widely-used, proprietary outcome measurement tool used by health professionals to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Pain subscore is reported ranging from 0 to 100.
Time Frame: Baseline and Week 52
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo
Number analyzed (Participants) | 112 | 117 | 110 | 116
score on a scale | -24.7 (2.5) | -29.0 (2.1) | -25.5 (2.1) | -26.7 (2.2)
Statistical Analysis 1: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.405, ANCOVA; Mean Difference (Final Values) = -2.38, 95% CI 2-sided [-8.00 to 3.24]
Statistical Analysis 2: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.552, ANCOVA; Mean Difference (Final Values) = 1.89, 95% CI 2-sided [-4.37 to 8.16]
Statistical Analysis 3: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.763, ANCOVA; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [-4.91 to 6.68]

9. Other Pre Specified Outcome: Change From Baseline OA Function in the Target Knee
Description: Change from baseline OA function in the target knee as assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Numeric Rating Scale (NRS 3.1) physical functioning subscore (WOMAC Function) at Week 52. The WOMAC is a widely-used, proprietary outcome measurement tool used by health professionals to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Function subscore is reported ranging from 0 to 100.
Time Frame: Baseline and Week 52
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo
Number analyzed (Participants) | 112 | 117 | 110 | 116
score on a scale | -24.1 (2.5) | -29.6 (2.0) | -24.9 (2.1) | -25.1 (2.3)
Statistical Analysis 1: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.173, ANCOVA; Mean Difference (Final Values) = -3.90, 95% CI 2-sided [-9.50 to 1.71]
Statistical Analysis 2: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.724, ANCOVA; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [-5.12 to 7.36]
Statistical Analysis 3: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.914, ANCOVA; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-6.17 to 5.53]

10. Other Pre Specified Outcome: Change From Baseline in Medial Joint Space Width of Target Knee
Description: Change from baseline in medial joint space width as documented by X-ray of the target knee at Week 52.
Time Frame: Baseline and Week 52
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo
Number analyzed (Participants) | 112 | 117 | 110 | 116
mm | -0.04 (0.06) | -0.09 (0.06) | -0.16 (0.07) | -0.14 (0.06)
Statistical Analysis 1: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.529, ANCOVA; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.12 to 0.24]
Statistical Analysis 2: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.259, ANCOVA; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.08 to 0.28]
Statistical Analysis 3: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.807, ANCOVA; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.21 to 0.16]

11. Other Pre Specified Outcome: Change From Baseline OA Pain in the Target Knee [Unilateral Symptomatic OA]
Description: as for outcome 8
Time Frame: Baseline and Week 52
Population: Subjects with unilateral symptomatic OA in the ITT Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo
Number analyzed (Participants) | 45 | 35 | 45 | 39
score on a scale | -28.6 (3.5) | -30.1 (3.2) | -26.6 (3.1) | -23.8 (3.4)
Statistical Analysis 1: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.049, ANCOVA; Mean Difference (Final Values) = -8.73, 95% CI 2-sided [-17.44 to -0.03]
Statistical Analysis 2: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.211, ANCOVA; Mean Difference (Final Values) = -6.03, 95% CI 2-sided [-15.49 to 3.43]
Statistical Analysis 3: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.254, ANCOVA; Mean Difference (Final Values) = -5.23, 95% CI 2-sided [-14.24 to 3.78]

12. Other Pre Specified Outcome: Change From Baseline OA Function in the Target Knee [Unilateral Symptomatic OA]
Description: as for outcome 9
Time Frame: Baseline and Week 52
Population: Subjects with unilateral symptomatic OA in the ITT Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo
Number analyzed (Participants) | 45 | 35 | 45 | 39
score on a scale | -29.0 (3.9) | -29.9 (3.4) | -25.6 (3.1) | -21.5 (3.8)
Statistical Analysis 1: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.036, ANCOVA; Mean Difference (Final Values) = -10.26, 95% CI 2-sided [-19.82 to -0.69]
Statistical Analysis 2: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.170, ANCOVA; Mean Difference (Final Values) = -7.07, 95% CI 2-sided [-17.18 to 3.05]
Statistical Analysis 3: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.171, ANCOVA; Mean Difference (Final Values) = -6.29, 95% CI 2-sided [-15.33 to 2.74]

13. Other Pre Specified Outcome: Change From Baseline in Medial Joint Space Width of Target Knee [Unilateral Symptomatic OA]
Description: Change from baseline in medial joint space width as documented by X-ray of the target knee at Week 52.
Time Frame: Baseline and Week 52
Population: Subjects with unilateral symptomatic OA in the ITT Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo
Number analyzed (Participants) | 45 | 35 | 45 | 39
mm | 0.03 (0.10) | 0.19 (0.12) | -0.22 (0.11) | -0.21 (0.12)
Statistical Analysis 1: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.021, ANCOVA; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [0.06 to 0.72]
Statistical Analysis 2: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.131, ANCOVA; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.07 to 0.55]
Statistical Analysis 3: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.789, ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.35 to 0.26]

ADVERSE EVENTS:
Time Frame: Data regarding treatment-emergent adverse events (TEAEs) was collected in this study. TEAEs are events that were not present prior to study medication injection or, if present prior to study medication injection, had worsened in severity. The reporting period for TEAEs started after the injection of study medication on Study Visit Day 1 through Week 52 (End of Study)/Early Termination.
Description: Safety Analyses Set: All participants who were exposed to SM04690 or placebo. Safety was assessed using the actual treatment.
Groups:
- Other: Single intra-articular injection of an unidentified dose of SM04690 or Placebo due to incorrectly performed dilution or documentation by a pharmacist.
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.23 mg SM04690 | Placebo | Other
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/114 | 0/104 | 0/108 | 0/15
Serious Adverse Events (participants affected / at risk) | 5/111 | 4/114 | 4/104 | 3/108 | 1/15
Other Adverse Events (participants affected / at risk) | 25/111 | 23/114 | 19/104 | 18/108 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.03 mg SM04690 (N=111) | 0.07 mg SM04690 (N=114) | 0.23 mg SM04690 (N=104) | Placebo (N=108) | Other (N=15)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelitis transverse (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.03 mg SM04690 (N=111) | 0.07 mg SM04690 (N=114) | 0.23 mg SM04690 (N=104) | Placebo (N=108) | Other (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (16) | 13 (14) | 9 (13) | 10 (12) | 4 (6)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased vibratory sense (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (6) | 2 (2) | 4 (4) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT02536833/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT02536833/SAP_001.pdf